CLINICAL TRIAL: NCT02464579
Title: Prospective Inquiry of Breastfeeding Success at the Department of Neonatology of University Hospital of Cologne and Analysis of Influencing Factors
Brief Title: Breastfeeding Rates at the Department of Neonatology of University Hospital Cologne
Acronym: BFRUHC
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Titus Keller, MD, Dr. med. Titus Keller, University Hospital of Cologne
Other Study IDs: UHC-N-15-013
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Newborn
Keywords: breastfeeding rate; preterm infant; neonatal intensive care unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to measure the breastfeeding success for all preterm and term newborns in our department of neonatology during the hospital stay and at the age of six months.

DETAILED DESCRIPTION:
A score was established which combines information on breastfeeding rate and breastmilk feeding rate, and used to monitor daily breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* Inborn or referred to our Department of Neonatology in the first week of life
* Informed consent of both parents or legal guardian

Exclusion Criteria:

* No informed consent of parent or legal guardian.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In-patients of the Department of Neonatology of Cologne.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-05-01; Primary Completion 2016-06-30 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Rate | 6 months
  A score was established wich combines informations on breastfeeding rate and breastmilk rate into one value. Of special interest was the score at discharge from the neonatologic center.

CONTACTS AND LOCATIONS:
Overall Officials: Titus Keller, MD, Principal Investigator — Neonatology at the University Hospital of Cologne
Locations (1):
- Neonatology at University Hospital of Cologne, Cologne, Germany